CLINICAL TRIAL: NCT06644040
Title: A Randomized, Open-Label, Active-Controlled, 3-Way, Incomplete Block, Crossover, Single Escalating Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of TeriQ Patch in Healthy Adult Female Participants
Brief Title: A Study of TeriQ Patch in Healthy Adult Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QuadMedicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QD-TRP-101
Record Dates: First submitted 2024-10-07; First posted 2024-10-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TeriQ Patch (Experimental)
  Interventions: Drug: TeriQ Patch
- Teribone Injection (Active Comparator)
  Interventions: Drug: Teribone Inj.
- Forteo Injection (Active Comparator)
  Interventions: Drug: Forteo Inj.

INTERVENTIONS:
Drug: TeriQ Patch — Participants will receive two single doses of either of the TeriQ patch (Strength- 28.2 µg, 56.5 µg, and 113.0 µg) approximately 1 week apart.
  Route of administration- Dermal patch
  Other Names: Study Drug
  Arms: TeriQ Patch
Drug: Teribone Inj. — Participants may receive either one single dose Teribone Inj. or Forteo Inj. following TeriQ patch.
  Route of administration: Sub-cutaneous Injection
  Other Names: Control Drug 1
  Arms: Teribone Injection
Drug: Forteo Inj. — Participants may receive either one single dose Teribone Inj. or Forteo Inj. following TeriQ patch.
  Route of administration: Sub-cutaneous Injection
  Other Names: Control Drug 2
  Arms: Forteo Injection

SUMMARY:
This will be a single center, open-label, active-controlled, 3-way, incomplete block, crossover, randomized, and single escalating dose study.

DETAILED DESCRIPTION:
This study will compare TeriQ Patch with two active comparators, Teribone Injection and Forteo Injection, to evaluate the safety, tolerability, and pharmacokinetics of TeriQ Patch in healthy adult female participants.

This study will be a single escalating dose study in which 24 healthy adult female participants will receive 2 of the 3 TeriQ Patch dose levels (28.2 μg, 56.5 μg, and 113.0 μg) and 1 of the control drugs (Teribone Inj. or Forteo Inj.) in 3 separate time periods. There will be a washout period of approximately 1 week between each treatment period. The control drug will be administered as a subcutaneous (SC) injection and the test drug will be administered as a dermal patch.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult females aged 18 to 60 years (inclusive) at the time of Screening.
2. Those who weigh ≥ 45 kg and have a calculated BMI of 18.0 to 32.0 kg/meter square
3. Females must be non-pregnant and non-lactating and must use an acceptable, highly effective method of contraception (as defined below) in the case of heterosexual intercourse. Participants in an exclusive same-sex relationship are not required to adhere to contraceptive requirements. (However, they must not attempt pregnancy with donor eggs/sperm):

   * For the female, established hormonal contraception (oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, hormonal intrauterine system (IUS), or the vaginal ring) with the use of a condom for the male partner from 30 days prior to dosing and for at least 90 days after the last IP administration.
   * For the female, an intrauterine device (IUD) placed 30 days prior to first dosing and for at least 90 days after the last IP administration, with the use of a condom for the male partner.
   * For the female, surgical sterilization (with documented evidence or verbal confirmation) at least 6 months prior to Screening (eg, bilateral tubal occlusion, complete hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, tubal ligation).
   * For the male partner, a vasectomy at least 90 days prior to enrollment (with appropriate post vasectomy documentation or verbal confirmation of the absence of sperm in semen), provided the male partner is a sole partner.
   * Women not of childbearing potential must be postmenopausal for ≥ 12 months. Postmenopausal status may be confirmed through testing of FSH levels ≥ 40 IU/L at Screening for amenorrheic female subjects, at the discretion of the Investigator, or subject considered to be of childbearing potential.
   * Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day -1 and be willing to have additional pregnancy tests as required throughout the study.
   * For the female, total abstinence from heterosexual intercourse, if this is their usual practice, for 30 days prior and for 90 days after the last study treatment is acceptable. Periodic abstinence (eg, calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable forms of contraception.
4. Those who have received and fully understand a detailed explanation of this study, voluntarily decide to participate, and agree in writing to comply with the precautions.

Exclusion Criteria:

1. Those who have or have had a history of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immune, dermatologic, neurologic, active chronic condition or psychiatric disorders.
2. Those who have an acute illness within 28 days (or shorter if deemed suitable at the discretion of the Investigator) of administration of the IMP.
3. Those who have a medical condition that may affect the absorption, distribution, metabolism, or excretion of drugs.
4. Those who have any of the following conditions:

   * Metabolic bone disease (including hyperparathyroidism and Paget's disease of the bone),
   * Previous radiation therapy history, or Patients with history of or current skeletal malignancies or bone metastases.
   * Chronic kidney disease, autoimmune disorders, systemic corticosteroid use, hyperparathyroidism and urinary stones.
5. Those who demonstrate any of the following results from laboratory tests (laboratory tests may be repeated once if deemed appropriate by the Investigator):

   * Corrected serum Ca concentration > 2.7mmol/L

     1. Serum albumin < 40 g/L: corrected using the following formula,
     2. Serum albumin ≥ 40 g/L: measured value will be deemed to be the corrected value,
     3. Corrected Ca: Measured Calcium [(measured Albumin- 41) *0.02]
   * Individuals with a calculated creatinine clearance of 80mL/min or less
   * Those whose creatinine clearance calculated with the Cockcroft-Gault formula is 80 mL/min or less
   * (Creatinine Clearance = (((1.23 x weight x (140 - age))/creatinine) x 0.85) [if female],
   * QTcF > 470 msec,
   * Increase of alkaline phosphatase (> 1.5 x ULN),
   * PTH > 2.65pmol/L with abnormal high corrected Ca (as defined above).
6. Subjects whose blood pressure measured at the Screening visit or at pre dose falls under the range below or subjects with orthostatic hypotension (ie, drop of 20 mmHg systolic or 10 mmHg diastolic blood pressure):

   * Systolic blood pressure: 100 mmHg or less or greater than 159 mmHg,
   * Diastolic blood pressure: 60 mmHg or less or greater than 99 mmHg. Blood pressure assessments may be repeated twice if deemed appropriate by the Investigator.
7. Those who used any prescription medications, within 14 days of IMP administration are excluded, however hormonal contraceptives are considered an exception.
8. Those who use any medical preparations (including over the counter [OTC] drugs, herbal medications, and nutritional and vitamin supplements within 7 days of IMP administration are excluded; however, short term, episodic use up to 4g daily paracetamol is permitted.
9. Those who are unable to eat clinic-provided standard meals. Specific dietary requirements (such as vegan/vegetarian options or halal alternatives) are acceptable at the discretion of the Investigator.
10. Those who have donated blood or plasma of approximately 500 mL within 90 days of the IMP administration, or those who have received a blood transfusion within 1 month prior to the date of administration.
11. Those who have participated in another clinical study or bioequivalence study within 30 days or 5 half-lives (whichever is longer) of the first dose date (date of last dose of IMP).
12. Those who consume excessive amounts of caffeine (ie, more than 5 cups of coffee or equivalent per day) and are unable to abstain from consumption of caffeine products during the study period.
13. Those who consume excessive amounts of alcohol (ie, more than 14 standard drinks per week) or those who are heavy smokers (consuming more than 5 cigarettes or equivalent per day) and are unable to abstain from consuming alcohol or tobacco products from 3 days prior to study drug administration and during the study.
14. Those who are deemed by the Investigator to be unsuitable for participation in the study due to laboratory test results or other reasons (e.g., failure to comply with requests and instructions, uncooperative behavior).
15. Those with tattoos or other skin marks or blemishes at the IP application site that may, in the opinion of the Investigator, interfere with the ability to perform a local assessment of skin reactions.
16. Those with a history of substance abuse or test positive for drugs of abuse (including tetrahydrocannabinol [THC], cocaine, amphetamines, barbiturates, benzodiazepines, opiates, methadone, methamphetamines, methylenedioxymethamphetamine [MDMA], and phencyclidine [PCP]) on a urine drug Screening test.
17. Pregnant women and nursing mothers.
18. Those who tested positive for HBsAg, HBcAb, anti-HCVAb, anti-HIVAb, and syphilis (VDRL).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Yes
Enrollment: 24 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- Maximum plasma concentration (Cmax) | 12 timepoints on baseline up to 8 hours post first dose administration
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- Time for maximum plasma concentration (Tmax) | 12 timepoints on baseline up to 8 hours post first dose administration
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- Area under curve (AUC) | 12 timepoints on baseline up to 8 hours post first dose administration
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- half life | 12 timepoints on baseline up to 8 hours post first dose administration
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- Clearance (CL/F) | 12 timepoints on baseline up to 8 hours post first dose administration
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- Volume distribution (Vd/F) | 12 timepoints on baseline up to 8 hours post first dose administration
To evaluate the pharmacokinetic (PK) endpoints of teriparatide following a single dose administration of TeriQ Patch- Mean residence rate (MRT) | 12 timepoints on baseline up to 8 hours post first dose administration

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of teriparatide by number of participants with treatment related adverse events (TEAEs) | Screening to approximately 4 weeks post first dose administration
Number of participants with abnormal laboratory values and/or adverse events that are related to treatment. | Screening to approximately 4 weeks post first dose administration
Number of participants with changes to local stimulus response rate. | 3 timepoints on baseline post first dose administration (predose, 4hours and 8 hours after dosing)
  Local stimulus response test will be performed for the following items (pain, redness, swelling, itching, and hardness) before each administration. (within 60 minutes) and 4 and 8 hours after administration.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Linear Clinical Research Ltd., Joondalup, Western Australia
  - Linear Clinical Research Ltd., Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No